CLINICAL TRIAL: NCT01681680
Title: Effect of Genetic Variation in the Transporter OCT2, MATE1 and MATE2-K on the Pharmacokinetics and Pharmacodynamics of Metformin
Brief Title: Effect of Genetic Variation in the Transporter OCT2, MATE1 and MATE2-K on the PKPD of Metformin
Acronym: #6112
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6112
Record Dates: First submitted 2012-08-01; First posted 2012-09-10 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Other): Subjects will be given an oral dose of metformin once per day for two days.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Subjects will be given an oral dose of metformin once per day for two days.
  Other Names: GLUCOPHAGE

SUMMARY:
The current study is part of a large multi-investigator grant to look at the pharmacogenetics of a number of membrane transporters. The investigators will study individuals with particular genotypes of the human organic cation transporter, (hOCT2), and the multidrug and toxin extrusion transporters, MATE1, MATE2-K to test the hypothesis that genetic variation in hOCT2, hMATEE1 and hMATE2-K are associated with variation in the pharmacokinetics and/or pharmacodynamics of the antidiabetic agent, metformin.

DETAILED DESCRIPTION:
In the proposed study, a genotype to phenotype strategy is employed to study the role of the transporters, OCT2, MATE1, and MATE2-K and related variants in response and disposition to a known substrate, metformin. Recently, one polymorphic variant in MATE1 (PMT4302, g.-66T>C) showed decreased promoter activity by 40-45% (p<0.01), and one MATE2-K variant (PMT5597, g.-130G>A) showed increased promoter activity by 30% (p<0.05), compared to the reference. Both are the most common promoter variants in each gene (the frequencies of PMT4302: 32.1% and 23.1% in Caucasian and Asian; PMT5597: 26.2% and 48.5% in Caucasian and Asian) (unpublished data, Giacomini group). Specifically, the investigators will measure renal clearance of metformin, and plasma glucose and insulin levels, in healthy Caucasian and Asian subjects who carry either the reference or variant alleles in order to evaluate the effects of these variants on metformin disposition and response.

ELIGIBILITY:
Inclusion Criteria:

* Subjects self-identify racial background, identify themselves, parents and four grandparents as Caucasian and or Chinese.
* Subject status is healthy volunteer from the SOPHIE cohort
* Subjects over 18 years old
* Subjects who are healthy on the basis of medical history, physical examinations and laboratory tests if healthy volunteer from SOPHIE
* Subjects who agree with the written informed consent to participate in the study.

Exclusion Criteria:

* Under 18 years old
* Pregnant or lactating woman (female subjects will have a urine pregnancy test at the Day 1 visit)
* They report a prior history of any allergic reaction to metformin
* Has a risk of congestive heart failure requiring pharmacologic treatment (medical history)
* Has a prior history of renal* or hepatic dysfunction (renal and hepatic function will be evaluated based on screening blood tests conducted prior to study enrollment)
* Anemic (screening lab values, hemoglobin <10 g)
* Taking a medication that could confound study results (such as known substrates or inhibitors of OCT2, MATE1 and MATE2-K such as cimetidine)
* Subjects are undergoing radiologic studies involving intravascular administration of iodinated contrast materials, because use of such products may result in acute alteration of renal function
* They do not consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Renal clearance of Metformin based on genotypes | Study day procedures 48 hours
  Renal clearance of Metformin of study participants using reference genotype for transporters of OCT2, MATE1, and MATE2-K. In addition, Cmax for plasma glucose will be analyzed for all study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Giacomini, PhD, Principal Investigator — University of California, San Francisco